CLINICAL TRIAL: NCT02273986
Title: Drug-Drug Interaction Study in Health Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Kowa Research Institute, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: K-877-106
Record Dates: First submitted 2014-10-22; First posted 2014-10-24 (Estimated); Last update posted 2014-10-24 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
Keywords: Adult Volunteers
MeSH Terms: interventions — Digoxin; K-877 compound

ARMS (2):
- Digoxin (Experimental): Digoxin
  Interventions: Drug: Digoxin
- Digoxin with K-877 (Experimental): Digoxin with K-877
  Interventions: Drug: Digoxin; Drug: K-877

INTERVENTIONS:
Drug: Digoxin
Drug: K-877
  Arms: Digoxin with K-877

SUMMARY:
The purpose of this study is to assess the effects of K-877 on the pharmacokinetics of digoxin in healthy adult volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Subject is a healthy adult male or female volunteer between the ages of 18 and 45 years, inclusive, at Screening.
* Subject has a body mass index of 18 to 30 kg/m2, inclusive, at Screening.
* Subject has hematology, serum chemistry, and urinalysis test results within the reference ranges or is showing no clinically relevant deviations, as judged by the investigator at Screening.

Exclusion Criteria:

* Subject has clinically relevant abnormalities in the screening or check in assessments.
* Subject has a blood pressure (as measured at Screening during the collection of vital signs) after resting supine for at least 5 minutes that is higher than 140 mm Hg systolic or 90 mm Hg diastolic, or lower than 90 mm Hg systolic or 60 mm Hg diastolic (for males) and 50 mm Hg diastolic (for females).
* Subject has a supine pulse rate (as measured at Screening during collection of vital signs) after resting for 5 minutes that is outside the range of 40 to 90 beats per minute.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2014-08; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Maximum concentration (Cmax) | 24 hours

SECONDARY OUTCOMES:
Area under concentration curve (AUC) | 24 hours

CONTACTS AND LOCATIONS:
Overall Officials: Stuart Campbell, Study Director — Kowa Research Institute, Inc.
Locations (1):
- PPD, Austin, Texas, United States